CLINICAL TRIAL: NCT00411125
Title: A Double-Blind, Double-Dummy, Randomized, Placebo-Controlled Crossover Phase I Study Assessing Pharmacokinetics and Pharmacodynamics of Two Different SMC021 0.8 mg Variants and the Effect of Timing of Drug Intake in Healthy Postmenopausal Women
Brief Title: Pharmacokinetics and Pharmacodynamics Study of Oral Salmon Calcitonin in Healthy Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CSMC021A2111
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Last update posted 2006-12-13 (Estimated); Status verified 2006-12

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Postmenopausal; osteoporosis; Pharmacokinetics/dynamics; Calcitonin
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — salmon calcitonin

INTERVENTIONS:
Drug: Oral salmon calcitonin

SUMMARY:
This is a phase I study to analyze bioavailability and pharmacodynamic of two different variants of oral salmon calcitonin (SMC021) in postmenopausal women

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal women

Exclusion Criteria:

* Previous treatment with other osteoporosis medication

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 40 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 86
Dates: Start 2006-08; Study Completion 2006-11

PRIMARY OUTCOMES:
Pharmacokinetic profile of the new variant compared to the current variant on Day 1
Effect on bone resorption biomarker on Day 1

SECONDARY OUTCOMES:
Effect on bone resorption biomarker 24 hours after the last dosing on Day 3
Effect on bone resorption biomarker after drug intake at different timepoints
Effect of dosing at different timepoints on the pharmacokinetic profile

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Basel, Study Director — Novartis Basel +41 61 324 1111
Locations (1):
- Copenhagen, Denmark

REFERENCES:
- [Derived] Karsdal MA, Byrjalsen I, Riis BJ, Christiansen C. Investigation of the diurnal variation in bone resorption for optimal drug delivery and efficacy in osteoporosis with oral calcitonin. BMC Clin Pharmacol. 2008 Dec 4;8:12. doi: 10.1186/1472-6904-8-12. PMID 19055791